CLINICAL TRIAL: NCT00630825
Title: The Effect of Dose Titration of LY2189265 in Overweight and Obese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Dose Titration of LY2189265 in Overweight Participants With Type 2 Diabetes Mellitus
Acronym: EGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12068; H9X-MC-GBCJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.0/2.0 milligram (mg) LY2189265 (Experimental): LY2189265: 1.0 milligram (mg), subcutaneous (SC) injection, once weekly (QW) for 4 weeks; followed by 2.0 mg, SC injection, QW for 12 weeks
  Interventions: Drug: LY2189265
- 1.0/1.0 milligram (mg) LY2189265 (Experimental): LY2189265: 1.0 mg, subcutaneous (SC) injection, once weekly (QW) for 16 weeks
  Interventions: Drug: LY2189265
- 0.5/1.0 milligram (mg) LY2189265 (Experimental): LY2189265: 0.5 milligram (mg), subcutaneous (SC) injection, once weekly (QW) for 4 weeks; followed by 1.0 mg, SC injection, QW for 12 weeks
  Interventions: Drug: LY2189265
- Placebo (Placebo Comparator): Placebo: subcutaneous (SC) injection, once weekly (QW) for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: 0.5/1.0 milligram (mg) LY2189265; 1.0/1.0 milligram (mg) LY2189265; 1.0/2.0 milligram (mg) LY2189265
Drug: Placebo
  Arms: Placebo

SUMMARY:
To study once weekly injections of LY2189265 compared to placebo on blood glucose by measuring glycosylated hemoglobin (HbA1c) change from baseline after 16 weeks in overweight Type 2 Diabetes Mellitus participants.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus >3 months by history prior to entering the trial, based on disease diagnostic criteria from the American Diabetes Association (ADA 2007).
* Men or women 18 years of age or older. Women must have a negative pregnancy test and be willing to use birth control during study duration and one month post.
* Have glycosylated hemoglobin (HbA1c) of >7.0% to ≤10.5% as determined by central laboratory at screening.
* Have a body mass index (BMI) between 27 and 40 kilograms/meter squared (kg/m^2), inclusive.
* Have been on the same doses for 3 months of any approved combination of 2 oral antihyperglycemic medications in any combination of the following: sulfonylureas (e.g. Chlorpropamide or Diabinese, Glimepiride or Amaryl, Tolbutamide or Orinase, Tolazamide or Tolinase, Glipizide or Glucotrol, Glyburide also known as Micronase, Diabeta, or Glynase), biguanides (e.g. Glucophage or metformin), thiazolidinediones (e.g. Rosiglitazone or Avandia, or Pioglitazone or Actos), or dipeptidyl peptidase 4 (DPP-IV) inhibitors (e.g. Sitagliptin or Januvia). A combination pill of any 2 of these drugs is allowed (1 only), (e.g. Metformin and Glipizide or Metaglip), (e.g. Metformin and Glyburide or Glucovance), (e.g. Pioglitazone and Glimepiride or Duetact), or (e.g. Sitagliptin and Metformin or Janumet).

Exclusion Criteria:

* Have known Type 1 Diabetes Mellitus
* Have taken glucagon-like peptide-1 (GLP-1) or any GLP-1 analog drug (Byetta)
* Have a history of unstable angina, heart attack (myocardial infarction), heart arrhythmia (ventricular), congestive heart failure, or other coronary intervention (percutaneous transluminal coronary angioplasty [PTCA], open heart surgery, or coronary artery bypass graft [CABG]), a transient ischemic attack (TIA) or stroke (cerebrovascular accident) in the last 6 months prior to screening.
* Have acute or chronic hepatitis or elevated liver function tests (alanine transaminase), a history of chronic or recurrent pancreatitis. Have renal disease or a serum creatinine (blood test) >2 milligrams per deciliter (mg/dL). If taking biguanides (e.g. metformin or Glucophage), or DPP-IV inhibitors (e.g. Sitagliptin or Januvia or Janumet), creatinine must be ≤1.5 mg/dL.
* Currently taking prescription or over the counter medications to prevent weight loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon-Fri 9AM-5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (31):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biddeford, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomfield Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flemington, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Menomonee Falls, Wisconsin
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toa Baja

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.0/1.0 Milligram (mg) LY2189265: LY2189265: 1.0 milligram (mg), subcutaneous (SC) injection, once weekly (QW) for 16 weeks
- Placebo: Placebo: subcutaneous (SC), once weekly (QW) for 16 weeks
Period: Overall Study
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Started | 65 | 65 | 66 | 66
Received at Least One Dose of Study Drug | 65 | 65 | 66 | 66
Completed | 56 | 58 | 58 | 60
Not Completed | 9 | 7 | 8 | 6
Not completed — Adverse Event | 4 | 4 | 3 | 1
Not completed — Entry Criteria Not Met | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of LY2189265 or Placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo | Total
Number analyzed (Participants) | 65 | 65 | 66 | 66 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.49 (11.28) | 57.46 (11.72) | 58.65 (11.69) | 55.96 (12.49) | 56.65 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 31 | 37 | 129
  Male | 34 | 35 | 35 | 29 | 133
Race/Ethnicity, Customized [Number; unit: participants]
  African | 4 | 6 | 5 | 4 | 19
  Caucasian | 36 | 39 | 40 | 36 | 151
  East Asian | 1 | 0 | 0 | 0 | 1
  Hispanic | 23 | 20 | 19 | 26 | 88
  Native American | 1 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 57 | 58 | 227
  Puerto Rico | 9 | 9 | 9 | 8 | 35
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.43 (0.99) | 8.25 (0.99) | 8.25 (0.89) | 8.05 (0.82) | 8.24 (0.93)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meters (kg/m^2) | 34.24 (4.11) | 33.85 (3.95) | 33.70 (4.11) | 33.89 (4.31) | 33.92 (4.10)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 98.60 (18.41) | 96.68 (16.51) | 94.76 (16.53) | 94.74 (15.21) | 96.18 (16.68)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 8.63 (6.92) | 8.13 (5.43) | 8.97 (7.62) | 7.48 (5.41) | 8.30 (6.41)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) in Overweight and Obese Participants With Type 2 Diabetes Mellitus
Description: Once weekly injections of LY2189265 (titrated and non-titrated doses) compared to placebo on blood glucose were evaluated. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusting for treatment, combination of oral medications, and baseline glycosylated hemoglobin (HbA1c).
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable glycosylated hemoglobin (HbA1c) data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 62 | 63 | 65 | 65
percentage of glycosylated hemoglobin | -1.52 (0.12) | -1.29 (0.12) | -1.28 (0.12) | -0.27 (0.12)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed

2. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Fasting blood glucose is a test to determine how much glucose (sugar) is in a blood sample after an overnight fast. Least Squares (LS) means of change were calculated using analysis of covariance (ANCOVA) adjusting for treatment, combination of oral medications, and baseline.
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable fasting blood glucose data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 51 | 52 | 48 | 53
millimoles per liter (mmol/L) | -2.64 (0.33) | -2.04 (0.34) | -2.09 (0.34) | -0.49 (0.32)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed

3. Secondary Outcome: Meal Test Glucose Excursion (Change in Blood Glucose to Test Meal)
Description: Glucose excursion in response to a standardized solid mixed meal test was evaluated at baseline (randomization) and at Week 16, or at early termination. Each of the 2 standardized meal tests required participants to fast starting at 2200 hours the night prior to the test. A standardized breakfast meal was provided to the participant (approximately 550 kilocalorie [Kcal], 103 grams [g] carbohydrates, 22 g protein, and 8.5 g fat) and was to be consumed within 15 minutes. Serial venous blood samples were taken at the start of the meal (fasting [0]) and 30, 60, 90, 120, and 180 minutes after the start of the meal. Least Squares (LS) means of change in mean glucose area under the curve excursion following a test meal were calculated adjusting for treatment, combination of oral medications, and baseline.
Time Frame: Baseline and 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable glucose excursion data.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)*minute
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 52 | 56 | 54 | 59
millimoles per liter (mmol/L)*minute
  Baseline (n=63, n=62, n=66, n=63) | 11.03 (5.02) | 11.12 (4.77) | 10.32 (4.93) | 10.76 (4.37)
  Week 16 (n=52, n=56, n=54, n=59) | 8.16 (4.58) | 9.92 (5.32) | 8.85 (4.94) | 10.94 (4.79)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at Week 16. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.047, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.025, ANCOVA — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Daily Mean Blood Glucose Values From the 8-point Self Monitored Blood Glucose (SMBG) Profiles
Description: Change from baseline in mean daily blood glucose values were measured using self-monitored blood glucose (SMBG) data collected at the following 8 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening meal; 2 hours post-evening meal; bedtime; and 2:00 am. The daily mean was calculated as the average of the 8 blood glucose values collected on a particular day. Least Squares (LS) means of change from baseline of the mean of the 8 time points (Daily Mean) were calculated using analysis of covariance (ANCOVA) adjusting for treatment, combination of oral medications, and baseline.
Time Frame: 2 separate days in the week preceding the Baseline, Week 4, Week 8, and Week 16 visits.
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable blood glucose (SMBG) data. For Week 16 data, last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 41 | 50 | 46 | 49
milligrams per deciliter (mg/dL)
  Week 4 (n=34, n=38, n=35, n=41) | -31.19 (5.85) | -35.94 (5.30) | -31.66 (5.36) | -8.10 (5.06)
  Week 8 (n=34, n=41, n=38, n=41) | -43.00 (5.88) | -40.68 (5.43) | -36.02 (5.35) | -14.58 (5.38)
  Week 16 (n=41, n=50, n=46, n=49) | -37.49 (5.89) | -41.79 (5.25) | -32.52 (5.40) | -8.67 (5.30)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at Week 4. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at Week 8. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 5: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 4]
Statistical Analysis 6: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 4]
Statistical Analysis 7: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Beta (β)-Cell Function and Insulin Sensitivity as Estimated by the Updated Homeostasis Model Assessment Method (HOMA2)
Description: Homeostasis Model Assessment tool (HOMA2) of β-cell function is a technique for estimating beta-cell function (HOMA2-%B) and insulin sensitivity (HOMA2-%S) using basal serum glucose, and c-peptide concentrations. A fasting blood glucose, c-peptide, and serum insulin level were drawn for purposes of this determination just prior to the mixed meal test.
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable HOMA2-%B or HOMA2-%S data.
Measure: Mean (Standard Deviation); unit: percentage of HOMA2
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 47
percentage of HOMA2
  HOMA2-%B | 45.61 (55.20) | 44.26 (93.89) | 39.20 (45.56) | 1.04 (41.12)
  HOMA2-%S | 3.58 (18.51) | -1.65 (17.19) | 0.46 (13.78) | 2.46 (12.23)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison of HOMA2-%B. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.904, ANCOVA — Treatment comparison of HOMA2-%S. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 5: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.138, ANCOVA; Treatment comparison of HOMA2-%S. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 6: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.729, ANCOVA — [p-value comment as in outcome 5, analysis 4]

6. Secondary Outcome: Percentage of Participants Achieving a Glycosylated Hemoglobin (HbA1c) of <7% or ≤6.5%
Description: Percentages of participants who achieved glycosylated hemoglobin (HbA1c) levels of <7% or ≤6.5% were analyzed with a logistic regression model with baseline, combination of oral medications, and treatment as factors included in the model.
Time Frame: Baseline and 4 and 8 and 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable glycosylated hemoglobin (HbA1c) data. For Week 16 data, last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Number; unit: percentage of participants
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 66
percentage of participants
  HbA1c levels <7.0%, Baseline | 3.1 | 4.6 | 1.5 | 4.5
  HbA1c levels ≤6.5%, Baseline | 0.0 | 1.5 | 0.0 | 0.0
  HbA1c levels <7.0%, Week 4 | 15.4 | 30.8 | 22.7 | 7.6
  HbA1c levels ≤6.5%, Week 4 | 4.6 | 7.7 | 3.0 | 1.5
  HbA1c levels <7%, Week 8 | 41.5 | 47.7 | 47.0 | 15.2
  HbA1c levels ≤6.5%, Week 8 | 20.0 | 26.2 | 18.2 | 1.5
  HbA1c levels <7%, Week 16 | 53.8 | 50.8 | 56.1 | 15.2
  HbA1c levels ≤6.5%, Week 16 | 32.3 | 32.3 | 33.3 | 4.5

7. Secondary Outcome: Change From Baseline in Body Weight
Description: LS means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusting for treatment, combination of oral medications, and baseline.
Time Frame: Baseline, 4, 8, and 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable body weight data. For Week 16 data, last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 63 | 63 | 65 | 65
kilograms (kg)
  4 weeks (n=63, n=63, n=65, n=65) | -1.28 (0.23) | -1.08 (0.23) | -0.50 (0.22) | -0.06 (0.22)
  8 weeks (n=61, n=60, n=63, n=64) | -2.12 (0.31) | -1.67 (0.32) | -1.39 (0.31) | -0.12 (0.31)
  16 weeks (n=63, n=63, n=65, n=65) | -2.51 (0.38) | -1.40 (0.38) | -1.58 (0.37) | -0.07 (0.38)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 4 weeks. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.113, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 8 weeks. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 5: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 7, analysis 4]
Statistical Analysis 6: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 7, analysis 4]
Statistical Analysis 7: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 16 weeks. P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 8: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 7, analysis 7]
Statistical Analysis 9: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 7, analysis 7]

8. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Mean change from baseline in waist circumference (a measure of central obesity).
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable waist circumference data. For Week 16 data, last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 59 | 60 | 63 | 60
centimeters (cm) | -1.92 (4.24) | -1.51 (4.56) | -1.33 (4.21) | 0.20 (3.40)
Statistical Analysis 1: Comparison: 1.0/2.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 2: Comparison: 1.0/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.028, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed
Statistical Analysis 3: Comparison: 0.5/1.0 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.047, ANCOVA — P-values ≤0.05 were considered significant. No adjustment for multiple comparisons was performed

9. Secondary Outcome: Nausea and Dyspepsia Measured by Visual Analog Scale
Description: Participants were asked to score nausea and dyspepsia (abdominal pain and bloating) on a scale of 0 (none) to 100 after the largest meal of the day.
Time Frame: One week before and one week after each of the Baseline and Week 4 and Week 8 and Week 16 visits
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable nausea or dyspepsia (abdominal pain and bloating) data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 66
units on a scale
  Nausea, Week before Baseline (n=52, 57, 61, 57) | 4.81 (10.50) | 3.56 (6.46) | 3.70 (5.76) | 3.35 (5.83)
  Nausea, Week after Baseline (n=42, 46, 50, 50) | 5.07 (8.58) | 3.85 (6.46) | 3.86 (5.96) | 2.25 (4.82)
  Ab pain, Week before Baseline (n=52, 57, 61, 57) | 5.66 (11.37) | 3.55 (9.14) | 4.04 (7.15) | 3.63 (6.58)
  Ab pain, Week after Baseline (n=42, 46, 50, 50) | 5.82 (9.41) | 4.89 (13.35) | 4.51 (8.60) | 2.86 (7.27)
  Bloating, Week before Baseline (n=52, 57, 61, 57) | 11.49 (16.80) | 8.11 (18.04) | 10.21 (15.32) | 9.30 (18.65)
  Bloating, Week after Baseline (n=42, 46, 50, 50) | 8.95 (12.90) | 10.10 (16.64) | 9.17 (15.61) | 8.42 (20.05)
  Nausea, Week before Week 4 (n=42, 55, 52, 59) | 6.74 (10.89) | 6.88 (11.47) | 7.97 (15.33) | 4.10 (7.32)
  Nausea, Week after Week 4 (n=49, 58, 59, 54) | 18.13 (24.52) | 12.28 (19.46) | 7.91 (12.39) | 4.10 (7.57)
  Ab pain, Week before Week 4 (n=42, 55, 52, 59) | 6.28 (9.53) | 7.74 (13.89) | 6.38 (11.13) | 4.45 (9.19)
  Ab pain, Week after Week 4 (n=49, 58, 59, 54) | 12.47 (20.44) | 9.31 (15.77) | 4.94 (8.89) | 4.59 (7.88)
  Bloating, Week before Week 4 (n=42, 55, 52, 59) | 13.56 (19.51) | 12.00 (19.17) | 9.95 (13.27) | 7.96 (15.77)
  Bloating, Week after Week 4 (n=49, 58, 59, 54) | 19.90 (25.61) | 13.40 (21.15) | 10.23 (13.88) | 8.40 (14.96)
  Nausea, Week before Week 8 (n=50, 51, 55, 58) | 10.90 (20.26) | 5.45 (10.63) | 7.39 (13.53) | 6.11 (12.59)
  Nausea, Week after Week 8 (n=50, 54, 54, 55) | 8.58 (12.88) | 5.57 (11.50) | 8.69 (13.41) | 5.30 (11.52)
  Ab pain, Week before Week 8 (n=50, 51, 55, 58) | 10.76 (19.06) | 5.76 (12.47) | 5.12 (9.01) | 6.65 (13.15)
  Ab pain, Week after Week 8 (n=50, 54, 54, 55) | 7.97 (14.72) | 6.87 (14.56) | 6.26 (11.93) | 6.38 (12.74)
  Bloating, Week before Week 8 (n=50, 51, 55, 58) | 17.65 (26.41) | 10.93 (17.92) | 11.58 (20.13) | 10.12 (19.20)
  Bloating, Week after Week 8 (n=50, 54, 54, 55) | 13.30 (18.66) | 11.18 (19.56) | 14.50 (20.95) | 10.34 (17.17)
  Nausea, Week before Week 16 (n=45, 49, 52, 54) | 9.68 (17.79) | 3.31 (5.53) | 6.36 (10.82) | 5.88 (14.41)
  Nausea, Week after Week 16 (n=45, 48, 49, 53) | 11.09 (17.62) | 5.73 (10.80) | 7.77 (12.25) | 3.40 (6.40)
  Ab pain, Week before Week 16 (n=45, 49, 52, 54) | 6.46 (9.48) | 5.68 (11.09) | 6.26 (12.89) | 6.17 (14.24)
  Ab pain, Week after Week 16 (n=45, 48, 49, 53) | 7.56 (14.28) | 5.99 (11.53) | 6.44 (12.58) | 5.19 (11.72)
  Bloating, Week before Week 16 (n=45, 49, 52, 54) | 12.57 (18.93) | 9.06 (16.78) | 12.26 (20.06) | 9.30 (18.60)
  Bloating, Week after Week 16 (n=45, 48, 49, 53) | 14.06 (20.46) | 11.11 (19.62) | 14.04 (22.26) | 8.84 (17.44)

10. Secondary Outcome: Change From Baseline in Gastroparesis Cardinal Symptom Index (GCSI) Scores
Description: Gastroparesis Cardinal Symptom Index (GCSI) is a participant-completed questionnaire designed to assess the severity of symptoms consistent with delayed gastric emptying (nausea/vomiting, abdominal bloating, and stomach fullness) at each study visit. GCSI scores ranged from 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, to 5=very severe.
Time Frame: Baseline and 4 and 8 and 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable Gastroparesis Cardinal Symptom Index (GCSI) questionnaire data. For Week 16 data, last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 66
units on a scale
  Stomach fullness, Week 4 (n=62, n=60, n=65, n=65) | 0.55 (1.51) | 0.57 (1.35) | 0.62 (1.26) | 0.35 (1.39)
  Stomach fullness, Week 8 (n=59, n=60, n=59, n=63) | 0.46 (1.65) | 0.30 (1.33) | 0.71 (1.54) | 0.25 (1.39)
  Stomach fullness, Week 16 (n=63, n=62, n=65, n=65) | 0.21 (1.58) | 0.27 (1.28) | 0.51 (1.34) | 0.15 (1.34)
  Bloating, Week 4 (n=62, n=60, n=65, n=65) | 0.35 (0.10) | 0.28 (0.93) | 0.19 (0.91) | 0.28 (0.84)
  Bloating, Week 8 (n=59, n=60, n=60, n=63) | 0.41 (1.34) | 0.13 (1.02) | 0.14 (1.32) | 0.18 (0.92)
  Bloating, Week 16 (n=63, n=62, n=65, n=65) | 0.02 (1.04) | 0.11 (0.94) | 0.32 (1.32) | 0.28 (0.86)
  Nausea/Vomiting, Week 4 (n=62, n=60, n=64, n=65) | 0.25 (0.71) | 0.19 (0.71) | 0.22 (0.52) | 0.03 (0.40)
  Nausea/Vomiting, Week 8 (n=59, n=60, n=60, n=63) | 0.46 (0.97) | 0.04 (0.64) | 0.28 (0.62) | 0.02 (0.39)
  Nausea/Vomiting, Week 16 (n=63, n=62, n=65, n=65) | 0.20 (0.64) | -0.01 (0.59) | 0.27 (0.48) | -0.01 (0.36)

11. Secondary Outcome: Number of Participants With a Hypoglycemic Event
Description: A documented hypoglycemic episode is defined as an event which is associated with a measured blood glucose of ≤70 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]), even if it was not associated with symptoms, signs, or treatment. A severe hypoglycemic episode is defined as an event with a measured blood glucose of <50mg/dL. Participant reports of hypoglycemic events were collected at the beginning of each visit starting at Baseline. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 4, 8, and 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo.
Measure: Number; unit: participants
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 66
participants
  Documented Hypoglycemic Event, Week 4 | 17 | 17 | 17 | 9
  Documented Hypoglycemic Event, Week 8 | 11 | 13 | 15 | 10
  Documented Hypoglycemic Event, Week 16 | 6 | 10 | 7 | 8
  Severe Hypoglycemic Event, Week 4 | 0 | 0 | 0 | 0
  Severe Hypoglycemic Event, Week 8 | 0 | 0 | 0 | 0
  Severe Hypoglycemic Event, Week 16 | 0 | 0 | 0 | 0

12. Secondary Outcome: Rate of Hypoglycemia Per 30 Days
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and/or symptoms of hypoglycemia (for example, sweating, shakiness, tachycardia, etc.) or a documented blood glucose (BG) concentration of ≤70 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]), even if it was not associated with symptoms, signs, or treatment. The rate is the average number of days out of 30 that a participant reported hypoglycemia. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo.
Measure: Mean (Standard Deviation); unit: events per participant per 30 days
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 66
events per participant per 30 days | 0.69 (1.29) | 0.80 (1.60) | 0.70 (1.18) | 0.24 (0.54)

13. Secondary Outcome: Change From Baseline in Lipids
Description: Lipids include total cholesterol, low-density lipoprotein (LDL)-cholesterol, high-density lipoprotein (HDL)-cholesterol, and triglycerides.
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable lipid data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Full Range); unit: millimoles per liter (mmol/L)
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 66
millimoles per liter (mmol/L)
  Cholesterol (n=61, n=60, n=60, n=62) | -0.34 [-3.44 to 2.28] | -0.05 [-1.37 to 2.69] | -0.09 [-2.18 to 4.77] | 0.18 [-1.91 to 2.56]
  LDL-Cholesterol (n=61, n=60, n=60, n=61) | -0.26 [-2.80 to 2.23] | -0.09 [-1.22 to 1.58] | -0.07 [-1.39 to 4.27] | 0.10 [-0.83 to 2.12]
  HDL-Cholesterol (n=61, n=60, n=60, n=61) | -0.02 [-0.33 to 0.41] | -0.02 [-0.37 to 0.54] | 0.00 [-0.26 to 0.23] | 0.00 [-0.24 to 0.26]
  Triglycerides (n=61, n=60, n=60, n=61) | -0.16 [-7.63 to 2.22] | -0.02 [-4.84 to 2.96] | -0.16 [-4.25 to 2.96] | 0.00 [-7.39 to 5.69]

14. Secondary Outcome: Participants Perception of Medication Effectiveness Using the Perceptions About Medications - Diabetes, Short Version (PAM-D-S) Questionnaire
Description: The Perceptions about Medications - Diabetes, Short Version (PAM-D-S) questionnaire consisted of: 2 items in which respondents were asked about their satisfaction with their diabetes medication over the past week using a 6-point scale ranging from 1 "completely dissatisfied" to 6 "completely satisfied"; 10 items in which respondents were asked about the effectiveness of their diabetes medications in the past week using a 4-point scale ranging from 1 "all of the time" to 4 "none of the time"; and 15 items asking respondents to indicate the frequency of physical side effects in the past week using a 4-point scale ranging from 1 "all of the time" to 4 "none of the time." These items were exploratory items taken from a Diabetes Medicines Survey and had not been validated as a scale. The percentage of participants that rated their general health as good or better are summarized.
Time Frame: Baseline and 4 and 8 and 16 weeks
Population: Participants in the per-protocol population with evaluable PAM-D-S questionnaire data. The per-protocol population consisted of participants who received at least one dose of study medication, had no significant protocol violations, completed the double-blind treatment phase, and were compliant with the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 55 | 58 | 59 | 58
percentage of participants
  Baseline | 72.7 | 87.0 | 87.5 | 89.1
  Week 4 | 83.3 | 90.2 | 87.5 | 87.0
  Week 8 | 82.9 | 90.5 | 90.9 | 88.6
  Week 16 | 92.1 | 90.2 | 86.0 | 93.0

15. Secondary Outcome: Validation of the Psychometric Properties of the Perceptions About Medications - Diabetes, Short Version (PAM-D-S) Questionnaire
Description: This purpose of this outcome measure was to validate the PAM-D-S questionnaire for future use. Please refer to Outcome Measure #14 for a description of the PAM-D-S questionnaire and results collected. A preliminary analysis indicated modifications to the questionnaire were required and further study is necessary to complete the validation. Therefore, the PAM-D-S questionnaire was not validated as a part of Study H9X-MC-GBCJ.
Time Frame: Baseline and 4 and 8 and 16 weeks
Population: The items in the Perceptions about Medications - Diabetes, Short Version (PAM-D-S) questionnaire were exploratory items taken from a Diabetes Medicines Survey and had not been validated as a scale. Therefore, no participants were analyzed for validation purposes.
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Pharmacokinetics (PK) of LY2189265 - Area Under the Concentration Time Curve (AUC)
Description: The population mean estimates and standard deviations were calculated for pharmacokinetic parameters (area under the concentration time curve [AUC] at steady state from time zero to 168 hours after study drug administration).
Time Frame: Time zero to 168 hours after study drug administration at 4, 8, and 16 weeks
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 concentration data.
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265
Number analyzed (Participants) | 58 | 175 | 59
nanograms*hour/milliliter (ng*h/mL) | 14587 (5674) | 7876 (3064) | 4488 (1746)

ADVERSE EVENTS:
Arm/Group | 1.0/2.0 Milligram (mg) LY2189265 | 1.0/1.0 Milligram (mg) LY2189265 | 0.5/1.0 Milligram (mg) LY2189265 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/65 | 2/65 | 3/66 | 1/66
Other Adverse Events (participants affected / at risk) | 41/65 | 35/65 | 40/66 | 36/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0/2.0 Milligram (mg) LY2189265 (N=65) | 1.0/1.0 Milligram (mg) LY2189265 (N=65) | 0.5/1.0 Milligram (mg) LY2189265 (N=66) | Placebo (N=66)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cryptogenic organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0/2.0 Milligram (mg) LY2189265 (N=65) | 1.0/1.0 Milligram (mg) LY2189265 (N=65) | 0.5/1.0 Milligram (mg) LY2189265 (N=66) | Placebo (N=66)
Abdominal distension (Gastrointestinal disorders) | 9 (9) | 5 (5) | 3 (3) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 2 (2) | 5 (5) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 3 (3) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3) | 6 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 4 (4) | 5 (5) | 5 (9)
Nausea (Gastrointestinal disorders) | 9 (10) | 11 (11) | 9 (13) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (9) | 1 (1) | 3 (5) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Early satiety (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 1 (3) | 3 (5) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days